CLINICAL TRIAL: NCT06262451
Title: Fecal Microbiota Transplant National Registry
Status: Enrolling by invitation | Type: Observational
Sponsor: University of California, San Francisco (Other)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Other Study IDs: 20-30182; 5R24AI118629 (NIH)
Record Dates: First submitted 2024-01-31; First posted 2024-02-16 (Actual); Last update posted 2025-06-10 (Actual); Status verified 2025-06

CONDITIONS: Fecal Microbiota Transplant
Keywords: FMT

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
A national data registry of patients receiving fecal microbiota transplantation (FMT) or other gut-related-microbiota products designed to prospectively assess short and long-term safety and effectiveness. Neonates will not be enrolled at any site for this study. The study data will derive from patient and donors past and present medical records, research records, and records about phone calls made as part of this research. The patient data will also be used from the records on visits.

ELIGIBILITY:
Recipient Inclusion Criteria :

* Ability to give informed consent
* Receiving FMT or other gut-related microbiota product within 90 days after providing consent
* Access to internet and/or telephone

Donor Inclusion Criteria:

* Ability to give informed consent
* Providing stool sample for FMT

Exclusion Criteria:

* Incarceration

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Participants will be eligible for participation regardless of age, race, ethnicity, or gender. Pediatric patients may participate if consent is given by a guardian.
Sampling Method: Probability Sample
Enrollment: 10 (Estimated)
Dates: Start 2023-10-20 (Actual); Primary Completion 2032-10 (Estimated); Study Completion 2032-10 (Estimated)

PRIMARY OUTCOMES:
To assess short-term and long-term safety of FMT and other gut-related-microbiota products | 10 years
  The safety of FMT is currently the greatest concern related to its use, and characterizing the safety of FMT and subsequent gut-related-microbiota products is the primary goal of the Registry. Short-term adverse events relate primarily to the method of delivery (e.g. colonoscopy) and to acute infections or other AEs from the donor fecal material and should be readily definable and quantifiable.The human-to-human transfer of feces may be associated with long-term health risks to the recipient because the gut microbiota is composed of many components that have not been characterized and can change over time in ways that cannot be currently predicted. It is imperative to determine if FMT leads to unintended development of serious conditions due to the transfer of gut microbiota. In addition to infections, the possibility that gut microbiota associated with a disease phenotype will be transplanted and result in chronic disease in recipients must be assessed.

SECONDARY OUTCOMES:
To characterize effectiveness of FMT and other gut-related-microbiota products. | 10 years
  Current information on the efficacy of FMT in treating clinical disease is restricted to case reports, case series, and one randomized trial in recurrent CDI. Furthermore, only short-term follow-up is generally provided in these reports. Determining the short-term and long-term effectiveness in real-world practice is crucial and assessing variations in efficacy outcomes related to methodology will enable standardization and optimization of FMT practice.
To gather information on FMT practice in North America | 10 years
  FMT and future methods of providing gut-related microbiota for treatment of disease are in their infancy. Currently there is a lack of standardization in all aspects of FMT, and given a lack of current regulatory requirements for reporting, the methodology being employed (e.g., screening, preparation, delivery, indications, follow-up) is unclear. Obtaining information on current FMT methods in North America is an important first step in characterizing FMT practice with the future goal of standardizing and optimizing FMT.
To promote scientific investigation. | 10 years
  A large FMT registry will provide an unprecedented and rich resource for investigators to advance the science of the gut microbiome in health and disease. The registry database will be available to investigators, with study proposals submitted for review by a Data Access and Publications Committee. Furthermore, this registry data will link to a biobank of fecal samples from the donor (one time) as well as recipient (before and after FMT). Together with the clinical metadata collected within the registry, information from analysis of specimens in the biobank will enhance short- and long-term safety surveillance as well as be a rich source of data to investigate modulation of the human gut microbiome.
To aid practitioners and sponsors in satisfying regulatory requirements | 10 years
  The FDA is currently determining the appropriate regulatory requirements for physicians performing FMT, exercising enforcement discretion regarding an IND requirements for use of FMT in treatment of CDI unresponsive to standard therapies. Participation in the FMT Registry provides an excellent method of oversight, helping to prevent marked departures in methodology from recommended practices, improve safety for patients, and gather data for quality improvement and future regulatory requirements. In addition, gut-related-microbiota products, from processed stool to defined microbiota consortia, require submission for regulatory approval. The Registry may function as an important vehicle for sponsors of gut-related microbiota products to satisfy pre-approval and post-approval assessment of product safety and efficacy.

CONTACTS AND LOCATIONS:
Overall Officials: Max Brondfield, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California, San Francisco, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No